CLINICAL TRIAL: NCT03156400
Title: Assessment of Autonomic Function and Cardiovascular Response to Exercise Testing in Parkinson's Disease Patients
Brief Title: Parkinson's Autonomic Responses to Treadmill Walking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Joseph Signorile, Professor, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20160709
Record Dates: First submitted 2017-03-03; First posted 2017-05-17 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Parkinson Disease; Autonomic Dysfunction
MeSH Terms: conditions — Parkinson Disease; Primary Dysautonomias | interventions — Exercise Test

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parkinson's disease (Active Comparator): Men and women can be included in the study if they are between 50 and 85 years of age and meet the following criteria:
  Have received clearance from a primary physician to perform a exercise stress test.
  Will be able to walk on a motorized treadmill with supporting harness system. Individual with PD who has recently had a diagnosis of Stage 1 or 2 on the Hoehn and Yahr scale.
  Interventions: Other: Exercise Stress Test
- Healthy Control (Active Comparator): Men and women can be included in the study if they are between 50 and 85 years of age and meet the following criteria:
  Have received clearance from a primary physician to perform a exercise stress test.
  Will be able to walk on a motorized treadmill with supporting harness system. Healthy individual with no unresolved cardiovascular, neuromuscular, and/or musculoskeletal disease.
  Interventions: Other: Exercise Stress Test

INTERVENTIONS:
Other: Exercise Stress Test — Gradual increase in treadmill grade while collecting respiratory gases.

SUMMARY:
This study will compare examine autonomic and cardiovascular responses to peak exercise testing in Parkinson's disease patients in varying stages of the disease, and healthy, age-matched participants. Participants will be asked to complete a peak exercise test on a motorized treadmill. Heart rate, blood pressure, norepinephrine, and other markers for cardiovascular function will be assessed at rest, during exercise, and post-exercise. The hypothesis to be tested is that Parkinson's disease patients will exhibit a decreased autonomic and cardiovascular response to exercise when compared to patients' healthy age-matched counterparts. The investigators secondary hypothesis is that Parkinson's disease patients in more advanced stages will exhibit a greater decrease in response when compared to these patients' Stage 1 counterparts, or healthy age-matched counterparts.

DETAILED DESCRIPTION:
This study will require the PD subjects to attend three testing days, lasting approximately 1 hour. PD subjects will report for two exercise testing sessions, with each session separated by 7 days. The age-matched, healthy subjects will only be required to attend two testing days consisting of one day for paperwork and anthropometric measurements, and one day for exercise testing, each lasting approximately 1 hour. PD subjects will be randomly assigned, in a counterbalanced manner, to either an "on-medication" or "off-medication" group for days two and three of testing. All subjects with PD will complete both exercise testing days.

Day 1: The subject will read and sign the informed and audio-visual consent forms and complete a health questionnaire, PAR-Q, and mini-mental survey. The subject will also complete the ACSM risk stratification screening questionnaire. Anthropometric measures will be taken to include, waist circumference, height, and weight. The subject will then be introduced to various test procedures which will be utilized throughout the experiment. Each subject will be familiarized with the treadmill and harness support system. The harness support system will be emplaced to ensure the safety of the PD patients due to the inherent fall risk associated with a progressive decline in motor control often seen in this population. The subject will walk on the treadmill at gradually increasing speeds until he or she indicates, by a prearranged signal, that a comfortable walking speed has been attained. Then the treadmill grade will be raised 2% every 30 seconds so the subject can feel what it is like to walk during a progressive test. This will last no longer than five minutes. PD subjects will also be given instruction as to which group (on, or off-medication) they have been assigned to, and how to prepare for the follow-on tests.

Off-Medication Testing Day: Subjects will complete a blood draw and a motorized treadmill VO2peak¬ test. Subjects are expected to arrive fasted (no food or drink for the past 12 hours) and having refrained from antiparkinsonian medication(s) for the past 24 hours. The subject will first be seated and given a 5 minute rest period. Following this rest period the phlebotomist will insert a catheter into the median cephalic vein in the antecubital (bend in the arm) region on the subject's arm. One vial (3 cc) of venous blood will be drawn prior to exercise testing and an identical draw will take place immediately following exercise testing. All blood specimens will be tested and analyzed at the University of Miami Miller School of Medicine. Then subject will then be allowed to eat a predetermined meal at the lab before returning to exercise. Following the meal, the subject will be asked to return to a seated resting position for an additional 5 minute period. During this time, gel electrodes will be applied on the subject for the purposes of ECG and heart/blood flow monitoring and measurements. Following this rest period, blood flow will be measured for an additional 5 minutes while the subject remains quietly seated. Next, the subject will be attached to the harness support system for the treadmill exercise test. For the metabolic assessment portion of the test, the subject will be fitted with a mask covering the nose and mouth, in which an airflow sensor will be attached to measure gas content during respirations. The test will start with a 4 minute warm-up at a speed dictated by the subject. By the end of the warm up, the subject will have reached a speed that both they and instructor agree upon which meets the requirements for moderate-intensity exercise. The speed will no longer be adjusted at this point. Percent grade will start at 2.5 percent and will be increased by 2.5 percent every 3 minutes until the subject has met the criterion for a peak exercise test, or has requested to stop. BP and HR will be monitored every minute of testing using an automatic electronic BP assessment machine (BPTRU, Coquitlam, BC), manual sphygmomanometer and stethoscope, and electronic ECG software (Cardiosoft, GE Healthcare), respectively. Successful completion of the test will be determined using the following criteria from the American College of Sports Medicine (ACSM): (1) plateau in VO2, (2) maximal HR within 10 beats per minute of an age predicted maximum, (3) a respiratory exchange ratio of >1.15, (4) respirations > 50 breaths per minute, (5) a rating of perceived exertion (RPE) ≥ 18. In addition to these criteria we will use ACSM indications for termination of an exercise test which include:

Absolute Indications

1. Suspicion of a myocardial infarction or acute myocardial infarction (heart attack)
2. Onset of moderate-to-severe angina (chest pain)
3. Signs of poor perfusion (circulation or blood flow), including pallor (pale appearance to the skin), cyanosis (bluish discoloration), or cold and clammy skin
4. Severe or unusual shortness of breath
5. Central Nervous System (CNS) symptoms e.g., ataxia (failure of muscular coordination), vertigo (an illusion of dizzying movement), visual or gait (pattern of walking or running) problems, confusion
6. Technical inability to monitor the ECG
7. Patient's request (to stop) Relative Indications

1. Any chest pain that is increasing 2. Physical or verbal manifestations of shortness of breath or severe fatigue 3. Wheezing 4. Leg cramps or intermittent claudication (grade 3 on a 4-point scale) 5. Hypertensive response (SBP >260 mm Hg; DBP>115 mm Hg) 6. Pronounced ECG changes from baseline (>2 mm of horizontal or down sloping ST- segment depression, or >2 mm of ST-segment elevation (except in aVR) 7. Exercise-induced bundle branch block that cannot be distinguished from ventricular tachycardia 8. Less serious arrhythmias (abnormal heart rhythms) such as supraventricular tachycardia On-Medication Testing Day: Procedures for the on-medication day will be identical to those used for the off-medication day testing. Each day, following the completion of exercise testing, subjects will be required to remain under lab personnel supervision until HR returns to within 10 beats of resting, and systolic BP returns to within 20 mmHg of resting. HR recovery will be measured continuously following exercise to determine how quickly it returns to baseline. This is a useful measure in determining autonomic function and the progression of PD symptoms.

ELIGIBILITY:
Inclusion Criteria:

Men and women can be included in the study if these potential participants are between 50 and 85 years of age and meet the following criteria:

* Have received clearance from a primary physician to perform a peak exercise test.
* Will be able to walk on a motorized treadmill with supporting harness system.
* Are Individuals with PD having recently had a diagnosis of Stage 1, or 2, or 3 on the Hoehn and Yahr scale and can present the research team with evidence from the potential participant's physician stating the diagnosis.

Or,

* The potential participant is a healthy individual with no unresolved cardiovascular, neuromuscular, and/or musculoskeletal disease.

Exclusion Criteria:

Men and women will be excluded from participation if the individual:

* Has been advised by a physician not to exercise.
* Is currently participating, or within the past 3 months has participated, in an exercise training program.
* Is currently on any cardiac or blood pressure medication.
* Has any additional neurological disorder.
* Is considered to be at high risk for cardiovascular disease as determined by the - American College of Sports Medicine (ACSM) risk stratification screening questionnaire or their primary physician.
* Is unable to provide informed consent.
* has a Mini-mental score less than 18.
* Is pregnant.
* Is currently a prisoner.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Blood Pressure Response | 12 minute
  Blood Pressure responses during increases in workload using automated blood pressure cuff
Cardiac Output using ergospirometry | 12 minute
  Cardiac responses during increases in workload using PhysioFlow automated respiratory gas ergospirometer
Vascular Resistance using ergospirometry | 12 minutes
  Changes in resistive force during increases in workload using PhysioFlow automated respiratory gas ergospirometer

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Signorile, PhD, Principal Investigator — University of Miami
Locations (1):
- Laboratory of Clinical Research, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No
IPD will be shared upon request from specific researchers